CLINICAL TRIAL: NCT02398214
Title: A Sleep Hygiene-based Intervention Program for Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201203083RIC
Record Dates: First submitted 2015-03-08; First posted 2015-03-25 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2016-10

CONDITIONS: Sleep
Keywords: Sleep; Infants; Toddlers; Behavioral intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep hygiene & standard care (Experimental): Participants receive a light, activity, and sleep training (LAST) intervention consists of behavioral and educational strategies for increasing light exposure and physical activity to minimize sleep disturbance.
  Interventions: Behavioral: Sleep hygiene
- Standard care (No Intervention): Participants receive usual care.

INTERVENTIONS:
Behavioral: Sleep hygiene — LAST intervention (light, activity, and sleep training) consists of behavioral and educational strategies for increasing light exposure and physical activity, minimizing television viewing and reducing television viewing time to < 2 hours per day, and engaging activities suitable to the child's motor development to minimize sleep disturbance.
  Arms: Sleep hygiene & standard care

SUMMARY:
Sleep problems during infancy are associated with behavior and emotional problems, poor language development , parental distress and mood disturbances, and overweight and obese children. The investigators proposed that children who receive the light, activity, and sleep training (LAST) intervention program in this study will have less parent report of problem sleep behaviors and longer duration of nighttime sleep compared to children with no intervention provided.

DETAILED DESCRIPTION:
Sleep problems are reported in 71.65% of our nation's infants and toddlers, and the prevalence is much higher than the 20-30% reported in Western countries. The investigators' preliminary findings also show that approximately 53-55% of parents of children between 6 and 12 months of age consider their child sleep a problem with about 4% not knowing whether their child sleep is a problem. Sleep development during infancy is characterized by increasing day-night differences in sleep-wakefulness such as longer bouts of sleep and fewer awakenings at night, and is driven by neurobiological maturation and environmental interactions. By 3 months of age, nearly 58% of infants can sleep continuously between 24:00-05:00 hours. When infants do not sleep through the night by 17 months of age, they are less likely to be able to do so at 29 months of age and beyond. Without proper intervention, sleep problems during infancy can persist to toddler and preschool age. Various interventions have been developed and tested in Western and Asian Countries to address the sleep problems in infants and young children, but none are in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton infant born at gestational age >= 37 weeks

Exclusion Criteria:

* Infants born before 37 weeks gestation
* Infants born with a congenital abnormality or a genetic disorder
* Parents with insufficient Chinese

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 247 (Actual)
Dates: Start 2012-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Actigraphic assessed sleep quantity variables | Baseline, 6-month follow-up, 12-month follow-up, and 18-month follow-up
  Total nighttime, daytime, and 24 hour sleep duration

SECONDARY OUTCOMES:
Actigraphic assessed sleep quality variables | Baseline, 6-month follow-up, 12-month follow-up, and 18-month follow-up
  Sleep onset latency and wake after sleep onset

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yu Tsai, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No